CLINICAL TRIAL: NCT05024279
Title: Pacing of the Left Bundle Branch Area NEcessitated After TAVR
Brief Title: Left Bundle Branch Area Pacing in Patients After TAVR
Acronym: PLANET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Moritz F. Sinner, Assistant Professor, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-0575
Record Dates: First submitted 2021-08-09; First posted 2021-08-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Aortic Valve Stenosis; AV Block; Pacing-Induced Cardiomyopathy
Keywords: left bundle branch area pacing; av block; right ventricular pacing; aortic valve stenosis; TAVR; ECG
MeSH Terms: conditions — Aortic Valve Stenosis; Atrioventricular Block

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Patients are randomized to receive left bundle branch are pacing due to higher degree AV block
  Interventions: Device: Left bundle branch area pacing
- Control Arm (Active Comparator): Patients are randomized to receive standard right ventricular pacing due to higher degree AV block.
  Interventions: Device: Right ventricular pacing

INTERVENTIONS:
Device: Left bundle branch area pacing — Left bundle branch area pacing will be applied as established in the literature using commercially available equipment.
  In case of unsuccessful application of left bundle branch area pacing, cross-over to right ventricular pacing is allowed.
  Arms: Intervention Arm
Device: Right ventricular pacing — Right ventricular pacing as the standard, established form of pacing will be applied in the control group. No cross-over to the intervention arm is anticipated.
  Arms: Control Arm

SUMMARY:
Prospective, randomized, single center clinical trial to compare the outcome of left bundle branch area pacing versus right ventricular apical pacing in patients with higher degree atrio-ventricular block and a normal left ventricular function after transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR) is a well-established treatment of aortic valve stenosis. Yet, requiry of permanent pacing due to new onset atrio-ventricular conduction block remains a frequent complication. Standard right ventricular pacing (RVP) at high pacing burden may lead to deterioration of left ventricular function. Left-Bundle-Area Pacing (LBBP) is a new, innovative method of physiological ventricular stimulation resulting in narrow, physiological QRS complexes.

In this prospective, randomized, single center clinica trial, patients are included after TAVR and with normal left ventricular function who require pacing due to a higher degree atriao-ventricular block with an anticipated high pacing burden. Patients will be randomized to receive either left bundle branch area pacing (intervention) or right ventricular apical pacing (control).

The results will confirm the feasibility of LBBP in patients following TAVR. Results will further investigate the primary outcome of a clinically relevant QRS narrowing and a combination of exploratory secondary endpoints including clinical outcomes, functional status, laboratory biomarkers, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Successful TAVR implantation for classical (high flow high gradient), symptomatic aortic valve stenosis
* LVEF ≥50%
* Guideline-based indication for pacing due to AV block III°, AV block II°, or symptomatic bradycardic atrial fibrillation with an expecteed ventricular pacing burden >20%
* Signed informeed conseent to study participation

Exclusion Criteria:

* LVEF <50%
* Expected pacing burden <20%
* Pre-existing implanted cardiac device
* Participation in a concurring interventional trial
* age <18 years
* Current preegnancy
* life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
QRS duration | 3 months
  QRS duration on 12-lead ECG, defined as earliest Q to latest S across all leads

SECONDARY OUTCOMES:
QRS duration | 12 months
  QRS duration on 12-lead ECG, defined as earliest Q to latest S across all leads
QRS duration | 24 months
  QRS duration on 12-lead ECG, defined as earliest Q to latest S across all leads
Death of any cause | 3 months
Death of any cause | 12 months
Death of any cause | 24 months
Death of cardio-vascular cause | 3 months
Death of cardio-vascular cause | 12 months
Death of cardio-vascular cause | 24 months
Re-hospitalization due to heart failure | 3 months
Re-hospitalization due to heart failure | 12 months
Re-hospitalization due to heart failure | 24 months
Change in left ventricular ejection fraction | 3 months
Change in left ventricular ejection fraction | 12 months
Change in left ventricular ejection fraction | 24 months
Change in echocardiographic left ventricular enddiastolic diameter | 3 months
Change in echocardiographic left ventricular enddiastolic diameter | 12 months
Change in echocardiographic left ventricular enddiastolic diameter | 24 months
Echocardiographic assessment of degreee of atrio-ventricular valve insufficiency | 3 months
Echocardiographic assessment of degreee of atrio-ventricular valve insufficiency | 12 months
Echocardiographic assessment of degreee of atrio-ventricular valve insufficiency | 24 months
Echocardiographic assessment of right ventricular ejection fraction | 3 months
Echocardiographic assessment of right ventricular ejection fraction | 12 months
Echocardiographic assessment of right ventricular ejection fraction | 24 months
Change in New York heart failure classification status | 3 months
Change in New York heart failure classification status | 12 months
Change in New York heart failure classification status | 24 months
Change in laboratory biomarkers NT-proBNP | 3 months
Change in laboratory biomarkers NT-proBNP | 12 months
Change in laboratory biomarkers NT-proBNP | 24 months
Change in functional status by 6 minute walk | 3 months
Change in functional status by 6 minute walk | 12 months
Change in functional status by 6 minute walk | 24 months
Change in EQ-5D quality of life | 3 months
Change in EQ-5D quality of life | 12 months
Change in EQ-5D quality of life | 24 months
Occurence of arrhythmias | 3 months
Occurence of arrhythmias | 12 months
Occurence of arrhythmias | 24 months

OTHER OUTCOMES:
Pacemaker-associated complications | 3 months
Pacemaker-associated complications | 12 months
Pacemaker-associated complications | 24 months
procedural implantation success | basline
  dichotomous yes / no
Implantation procedure duration | baseline
Fluoroscopy duration | baseline
Fluoroscopy dose | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Moritz F Sinner, MD, MPH, Principal Investigator — LMU Klinikum, Dept. of Cardiology; Stephanie Fichtner, MD, Principal Investigator — LMU Klinikum, Dept. of Cardiology
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No